CLINICAL TRIAL: NCT02186210
Title: Effect of Prewarming on Microcirculatory Response
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Prewarming_OPCAB
Record Dates: First submitted 2014-07-04; First posted 2014-07-10 (Estimated); Results first posted 2018-10-29 (Actual); Last update posted 2019-03-18 (Actual); Status verified 2014-08

CONDITIONS: Coronary Artery Bypass Graft Triple Vessel
Keywords: microcirculation; off-pump coronary artery bypass surgery; tissue oxygen saturation; vascular occlusion test; recovery slope

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- prewarming (Experimental): prewarming during induction of anesthesia
  Interventions: Device: prewarming
- control (No Intervention): no prewarming during induction of anesthesia

INTERVENTIONS:
Device: prewarming — recovery slope StO2
  Other Names: prewarming by active air heater
  Arms: prewarming

SUMMARY:
Intraoperative hypothermia may affect tissue microcirculation and can induce myocardial injury, wound infection, and coagulopathy. During off-pump coronary artery bypass surgery without cardiopulmonary bypass or induced hypothermia, maintenance of normothermia is important for clinical outcome. The investigators hypothesized that prewarming during induction of general anesthesia would reduce drop of body temperature and change of peripheral microcirculation.

DETAILED DESCRIPTION:
Microcirculatory parameters can be obtained from vascular occlusion test. Among those parameters, recovery slope during vascular occlusion test is known to reflect recruitment of microvasculature in response to hypoxic or ischemic insult. In this study, we will compare the recovery slope during vascular occlusion test between prewarming treatment group and control group.

ELIGIBILITY:
Inclusion Criteria:

* off-pump coronary artery bypass surgery

Exclusion Criteria:

* refuse to enroll
* cannot undergo vascular occlusion test: anatomical abnormality of both arms, severe peripheral vascular disease, presence of A-V fistula
* preoperative left ventricular ejection fraction < 35%
* preoperative continuous infusion of vasopressor or inotropes
* pregnancy

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2014-07; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yunseok Jeon, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cho YJ, Lee SY, Kim TK, Hong DM, Jeon Y. Effect of Prewarming during Induction of Anesthesia on Microvascular Reactivity in Patients Undergoing Off-Pump Coronary Artery Bypass Surgery: A Randomized Clinical Trial. PLoS One. 2016 Jul 21;11(7):e0159772. doi: 10.1371/journal.pone.0159772. eCollection 2016. PMID 27442052

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Prewarming | Control
Started | 20 | 20
Completed | 20 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Prewarming | Control | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 63 (9) | 66 (8) | 65 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 4 | 10
  Male | 14 | 16 | 30
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Korea, Republic of | 20 | 20 | 40

OUTCOME MEASURES:

1. Primary Outcome: Recovery Slope
Description: We will compare recovery slope assessed 3 hours after induction of anesthesia to evaluate the effect of prewarming during induction of anesthesia on microcirculation.
Time Frame: 3 hours after induction of anesthesia
Measure: Mean (Standard Deviation); unit: % / sec (recovery slope unit)
Arm/Group | Prewarming | Control
Number analyzed (Participants) | 20 | 20
% / sec (recovery slope unit) | 2.8 (1.0) | 3.1 (1.5)

2. Secondary Outcome: Tissue Oxygen Saturation
Time Frame: During the surgery, an average of 4 hours
Measure: Mean (Standard Deviation); unit: % (percent of tissue saturation)
Groups:
- Prewarming: prewarming during induction of anesthesia at 3 hr after induction
- Control: no prewarming during induction of anesthesia at 3 hr after induction
Arm/Group | Prewarming | Control
Number analyzed (Participants) | 20 | 20
% (percent of tissue saturation) | 76 (10) | 79 (7)

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Prewarming | Control
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes